CLINICAL TRIAL: NCT02108808
Title: Differential Effect of Ticagrelor vs Prasugrel or Clopidogrel Loading on Fractional Flow Reserve
Brief Title: Effect of Ticagrelor on Fractional Flow Reserve
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRAS CARDIOLOGY 18
Record Dates: First submitted 2014-04-04; First posted 2014-04-09 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Fractional Flow Reserve
Keywords: FFR; adenosine; Ticagrelor
MeSH Terms: interventions — Ticagrelor; Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel or Clopidogrel (Active Comparator): Prasugrel 60mg or Clopidogrel 600mg loading dose, as clinically indicated
  Interventions: Drug: Prasugrel or Clopidogrel
- Ticagrelor (Experimental): Ticagrelor 180mg loading dose
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor
  Arms: Ticagrelor
Drug: Prasugrel or Clopidogrel
  Arms: Prasugrel or Clopidogrel

SUMMARY:
Fractional flow reserve (FFR) is an established invasive method for assessing the physiological significance of coronary artery stenosis. Adenosine, an important endogenous regulator of coronary blood flow during both stress and ischemia, is widely used to achieve conditions of stable hyperemia required for measurement of FFR.

Studies in healthy volunteers and in patients with acute coronary syndrome (ACS) post percutaneous coronary intervention (PCI) receiving ticagrelor revealed a differential coronary blood flow velocity response during increasing doses of adenosine compared to placebo or prasugrel treated subjects, respectively. It has also been demonstrated that patients treated with ticagrelor have increased plasma adenosine levels. Therefore, it has been hypothesized that the degree of hyperemia obtained with adenosine infusion may be greater in patients on ticagrelor than that obtained in patients taking clopidogrel or prasugrel. If this proves to be true, it would lead to a lower FFR value with possible important clinical implications in ticagrelor receiving patients in need for FFR measurement.

This is a prospective, single center, randomized study of parallel design. Consecutive ticagrelor naive patients who are referred for coronary angiography and have an angiographically moderate to severe de novo stenosis (>50% and <90% diameter by visual assessment) in at least one major epicardial coronary artery amenable to PCI are candidates for this study. Patients after informed consent will be randomized (hour 0) to receive immediately post FFR (with adenosine iintravenous infusion at 140 μg/Kg/min for a 3 minute period) either ticagrelor 180mg loading dose or prasugrel 60mg/clopidogrel 600mg loading dose (as clinically indicated). FFR examination will be repeated 2 hours post loading dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Patients subjected to clinically indicated coronary angiography with at least one 50%-90% stenosis at 1 major epicardial vessel (by visual assessment) amenable to percutaneous coronary intervention.
3. Ticagrelor naive patients
4. Written informed consent

Exclusion Criteria:

1. History of coronary artery bypass surgery
2. Acute myocardial infarction within the previous 5 days
3. Known allergy to adenosine, ticagrelor, prasugrel or clopidogrel
4. Prior intracranial hemorrhage
5. Hemodialysis or creatinine clearance < 30ml/h
6. Moderate/severe hepatic failure
7. Active bleeding, or at increased risk of bleeding
8. Left ventricular ejection fraction <40%
9. Primary myocardial or valvular disease
10. Contraindication to adenosine
11. Angiographically visible thrombus at a target lesion, extremely tortuous coronary arteries, severely calcified lesions, left main disease, anatomy suitable for coronary artery bypass surgery
12. Previous q wave myocardial infarction in the area of target vessel
13. Severe left ventricular hypertrophy
14. Severe valvular heart disease
15. Heart failure as defined by New York Heart Association class III or IV 16.Hypotension (blood pressure <90 mm Hg)

17.Significant arrhythmia (e.g. excessive premature ventricular contractions or atrial fibrillation), tachycardia (heart rate >120 beats/min), bradycardia (<50 beats/min), increased risk for bradycardia 18.Caffeine consumption or cigarette smoking within the previous 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
% relative change in steady hyperemia FFR (sFFR) | 2 hours
  Steady hyperemia FFR (sFFR) is defined as the FFR value attained during stable hyperemia (as assessed by offline visual inspection of the 3-min hemodynamic trace) (sFFR post drug - sFFR pre drug)*100/sFFR pre drug between the 2 treatment arms

SECONDARY OUTCOMES:
% relative change in peak hyperemia FFR (pFFR) | 2 hours
  Peak hyperemia FFR is defined as the lowest FFR measurement during the first 60 sec of adenosine infusion (pFFR post drug - pFFR pre drug)*100/pFFR pre drug between the 2 treatment arms
% relative change in lowest FFR (lFFR) | 2 hours
  Lowest FFR (lFFR) is defined as the value provided by the automated FFR console (lFFR post drug - lFFR pre drug)*100/lFFR pre drug between the 2 treatment arms
% relative change in time to peak FFR (in seconds) | 2 hours
  (time to pFFR post drug - time to pFFR pre drug)*100/time to pFFR pre drug between the 2 treatment arms
% relative change in time to lowest FFR | 2 hours
  (time to lFFR post drug - time to lFFR pre drug)*100/time to lFFR pre drug between the 2 treatment arms
% relative change in area under the curve (AUC) of the FFR trace | 2 hours
  (AUC FFR post drug - AUC FFR pre drug)*100/AUC FFR pre drug between the 2 treatment arms

OTHER OUTCOMES:
Reclassification of coronary revascularization strategy at hour 2 in relation to hour 0 | 2 hours
  Number of patients who were reclassified regarding revascularization strategy at hour 2 in relation to hour 0, between the 2 treatment arms

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Achaia, Greece